CLINICAL TRIAL: NCT03323840
Title: Pilot for a Community Pharmacy Service Model: Impact of a Pharmacist Monitored Patient Blood Pressure Readings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20011451
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incentivized Care (Experimental): Patients will meet with the pharmacist up to 2 times/month for blood pressure measurement. Patients will receive a $10 gift card for each measurement.
  Interventions: Other: Incentivized Care

INTERVENTIONS:
Other: Incentivized Care — Patients will receive a $10 gift card for every blood pressure measurement (up to 2 times/month)

SUMMARY:
This study is designed to explore whether routine measurement of blood pressure by community pharmacists can improve patient adherence to blood pressure medications. The study will utilize an incentivized care approach, in which patients receive a $10 gift card for every time they come to the pharmacy for blood pressure management (up to 2 times/month). The investigators hypothesize that the simple process of coming in for a blood pressure measurement (without any other scripted interventions, counseling, or consultation) will be feasible and sufficient to improve adherence to medications. The investigators will also collect preliminary data to help estimate how these hypothetical improvements in adherence might result in improved blood pressure control, fewer office visits, and (ultimately) fewer adverse cardiovascular outcomes (i.e. heart attacks, strokes, etc).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of hypertension
* Current prescription for ≥2 antihypertensive medications for primary diagnosis of hypertension
* Prior use of ≥1 antihypertensive medication for ≥6 months at the same Kroger's Pharmacy (#523)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Age <18 years
* New diagnosis of hypertension within the prior 6 months
* Current pregnancy or lactation
* Limited English Proficiency
* Use of antihypertensive medications for secondary prevention of cardiovascular events. Patients with history of acute myocardial infarction, stroke, heart failure will be excluded, however, patients with diabetes will be eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Percentage of blood pressure measurements completed

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No